CLINICAL TRIAL: NCT07281053
Title: Use of Extended Platelet-Rich Fibrin Membranes in Comparison to Collagen Membranes for Socket Grafting: Part 2: A Randomized Clinical Trial
Brief Title: E-PRF vs Collagen Membranes in Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Advanced Rejuvenation and Esthetics (Network)
Responsible Party: Principal Investigator, Nathan Estrin, Periodontist, Center for Advanced Rejuvenation and Esthetics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13180-NEstrin
Record Dates: First submitted 2025-11-08; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Ridge Preservation
Keywords: Ridge preservation; extended platelet-rich fibrin; platelet-rich fibrin; Albumin-PRF

STUDY DESIGN:
Intervention Model Description: This research will be a 6-month randomized and controlled trial involving patients requiring at least one extraction and replacement with a dental implant. Participants will be recruited and randomly allocated to receive either one of the four iterations of using e-PRF membranes or a standard resorbable collagen membrane. All patients will be treated surgically with ridge preservation and dental implant placement using standard bone graft material and one of the membranes determined by their assigned group. Primary outcome includes radiographic ridge dimensions, soft tissue thickness, and wound healing outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not know which treatment they are receiving, Radiologist does not know which group recieved which treatment, and 3 blinded-clinicians will give wound healing scores according to Landy index
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Collagen Membrane (Active Comparator): Control group, Collagen membrane
  Interventions: Procedure: Barrier membrane for ridge preservation
- E-PRF membrane fabricated extra-orally (Experimental): E-PRF membrane fabricated extra-orally
  Interventions: Procedure: Barrier membrane for ridge preservation
- membrane w/solid (Experimental): E-PRF membrane fabricated extra-orally with a solid membrane overtop
  Interventions: Procedure: Barrier membrane for ridge preservation
- Bio-Filler (Experimental): E-PRF fabricated intra-orally as a Bio-Filler
  Interventions: Procedure: Barrier membrane for ridge preservation
- Bio-Filler w/solid (Experimental): E-PRF fabricated intra-orally as a Bio-Filler with a solid-PRF membrane overtop
  Interventions: Procedure: Barrier membrane for ridge preservation

INTERVENTIONS:
Procedure: Barrier membrane for ridge preservation — Various membranes utilized in ridge preservation were studied

SUMMARY:
Dental implants are often considered the gold standard to replace missing teeth. Having success with dental implants depends on the hard tissue and soft tissue remaining after tooth extractions. The first step to successful dental implant placement begins with proper socket grafting which includes placing a bone graft and membrane among other biomaterials such as platelet-rich fibrin (PRF) to prevent the collapse of the ridge that occurs after a dental extraction.

While platelet-rich fibrin is commonly utilized for ridge preservation, it is often used in conjunction with a collagen membrane due to the fact that it has a short resorption time lasting roughly 2 weeks. However, recently, it was discovered that by heating the plasma layer and denaturing the albumin, the resorption properties of PRF could be extended from 2 weeks to 4-6 months. This extended platelet-rich fibrin (e-PRF) membrane is a promising replacement to collagen membranes in various surgeries. The investigators previously demonstrated that e-PRF is a safe and feasible alternative to conventional membranes with 4 different iterations of applying the novel e-PRF membrane. However, there still lacks a comparative study to traditional collagen membranes and between the 4 different iterations.

Four different techniques utilizing e-PRF membranes for ridge augmentation will be performed with a collagen membrane as a control group. These techniques include 1) e-PRF as a sole barrier membrane, 2) layering a solid-PRF membrane over the e-PRF membrane, 3) fabricating e-PRF intra-orally in gel form as a Bio-Filler, and 4) Fabricating the e-PRF membrane intra-orally under a solid-PRF membrane.

DETAILED DESCRIPTION:
Dental implants are often considered the gold standard to replace missing teeth. Having success with dental implants depends on the hard tissue and soft tissue remaining after tooth extractions. The first step to successful dental implant placement begins with proper socket grafting which includes placing a bone graft and membrane among other biomaterials such as platelet-rich fibrin (PRF) to prevent the collapse of the ridge that occurs after a dental extraction.

While platelet-rich fibrin is commonly utilized for ridge preservation, it is often used in conjunction with a collagen membrane due to the fact that it has a short resorption time lasting roughly 2 weeks. However, recently, it was discovered that by heating the plasma layer and denaturing the albumin, the resorption properties of PRF could be extended from 2 weeks to 4-6 months. This extended platelet-rich fibrin (e-PRF) membrane is a promising replacement to collagen membranes in various surgeries. Previously, it was demonstrated that it is a safe a feasible alternative to conventional membranes with 4 different iterations of applying the novel e-PRF membrane. However, there still lacks a comparative study to traditional collagen membranes and between the 4 different iterations.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects requiring at least one extraction and replacement with a dental implant.
* No contraindications to dental implant placement

Exclusion Criteria:

* Smokers
* Autoimmune disease or disorder
* Neurologic disease or disorder
* Major mechanical obstruction to the mouth opening
* Acute capsulitis
* Bone metabolic disease
* Current systemic antibiotic treatment or within 3 months prior to the study
* Drug addiction or alcohol abuse
* Pregnancy, planning to become pregnant and or nursing
* Type 1 diabetes Uncontrolled Type 2 diabetes (Anyone with an A1c >= 7%)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Radiographic Vertical and Horizontal Dimensions measured in mm | 3 months
  Cone Beam Computed Tomography (CBCT) scans were acquired for all participants immediately after socket grafting and again at three months post-operatively. Horizontal ridge width was measured on cross-sectional images at three standard-ized apical levels relative to the alveolar crest: 1 mm (RW-1), 3 mm (RW-3), and 5 mm (RW-5). Measurements were conducted perpendicular to a vertical reference line drawn through the midpoint of the grafted socket. Buccal height (BH) and lingual height (LH) were measured at both time points as the linear distance from the most apical portion of the socket to the most coronal portion of the alveolar ridge, parallel to the same vertical reference line. Baseline buccal bone thickness (BBT) was measured on cross-sectional images at 1mm (BBT-1), 3mm (BBT-3), and 5mm (BBT-5) from the crest, parallel to a horizontal reference line.

SECONDARY OUTCOMES:
Soft tissue thickness measured in mm. | 3 months
  Soft tissue thickness was measured utilizing a standardized mechanical probing procedure with a #40 endodontic reamer equipped with an adjustable rubber stopper. Measurements were taken at the buccal crest, and 5 mm apical to the crest, both pre-operatively and at three months post-operatively, corresponding to the time of im-plant placement. Moreover, mid-occlusal soft tissue thickness (OSTT) was assessed at the three-month follow-up.
  At each measurement point, the reamer was gently advanced perpendicularly through the mucosa until hard tissue contact was obtained. The distance from the tip of the reamer to the rubber stopper was then calculated utilizing a digital caliper to identify soft tissue thickness. All measurements were carried out by a calibrated investigator under consistent positioning and lighting conditions to minimize variability.
Clinician reported wound healing outcomes | 2 weeks
  At the two-week post-operative visit, intraoral photographs of each extraction site were taken using a CANON digital camera. The images were independently assessed by three blinded clinicians utilizing the Landry, Turnbull, and Howley Wound Healing Index (LWHI). Healing was scored on a scale from 1 to 5, where 1 indicated very poor healing and 5 indicated excellent healing.
Time for membrane fabrication measured in seconds | intra-operative time.
  For all patients in the treatment groups, the time to fabricate and apply the e-PRF iteration was recorded. This included the time to draw blood into the collection tubes, centrifugation, using the Bio-Heat to denature albumin, cooling the tubes, mixing the e-PRF with liquid-PRF, allowing the membrane to set, harvesting and flattening the solid-PRF membranes, and intraoral application of the membranes.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakewood Ranch Dental, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Data will be provided to researchers conducting a meta-analysis.

DOCUMENTS (2):
  • Study Protocol (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT07281053/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT07281053/SAP_001.pdf